CLINICAL TRIAL: NCT06846671
Title: A Phase 3, Open-Label, Randomized Study of BGB-16673 Compared to Investigator's Choice (Idelalisib Plus Rituximab or Bendamustine Plus Rituximab or Venetoclax Plus Rituximab Retreatment) in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Previously Exposed to Both BTK and BCL2 Inhibitors
Brief Title: A Study of BGB-16673 Compared to Investigator's Choice in Participants With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Previously Exposed to Both Bruton Tyrosine Kinase (BTK) and B-cell Leukemia/Lymphoma 2 Protein (BCL2) Inhibitors
Acronym: CaDAnCe-302
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-302; 2024-518893-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: CLL; Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; idelalisib; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: BGB-16673 monotherapy (Experimental): Participants will receive BGB-16673 once daily until any of the treatment discontinuation criteria are met
  Interventions: Drug: BGB-16673
- Arm B: Investigator's Choice (Active Comparator): Participants will receive investigator's choice of idelalisib plus rituximab for CLL only or bendamustine plus rituximab, or venetoclax plus rituximab retreatment.
  Interventions: Drug: Bendamustine; Drug: Idelalisib; Drug: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: BGB-16673 — Administered orally
  Arms: Arm A: BGB-16673 monotherapy
Drug: Bendamustine — Administered intravenously
  Arms: Arm B: Investigator's Choice
Drug: Idelalisib — Administered orally
  Arms: Arm B: Investigator's Choice
Drug: Rituximab — Administered intravenously
  Arms: Arm B: Investigator's Choice
Drug: Venetoclax — Administered orally
  Arms: Arm B: Investigator's Choice

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of BGB-16673 compared with investigator's choice (idelalisib plus rituximab [for CLL only] or bendamustine plus rituximab or venetoclax plus rituximab retreatment) in participants with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) previously exposed to both BTK inhibitors (BTKi) and BCL2 inhibitors (BCL2i).

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia is a type of blood cancer that affects people around the world. People with CLL suffer from enlarged lymph nodes, spleen, or liver, or have symptoms like night sweats, weight loss and fever. They have shorter life expectancy compared to healthy people. There is an urgent need for new treatment to prolong life and control disease-related symptoms.

In this study, participants with relapsed/refractory (R/R) CLL who were previously exposed to a BTKi and a BCL2i will receive BGB-16673 or the investigator's choice of idelalisib plus rituximab (for CLL only) or bendamustine plus rituximab or venetoclax plus rituximab retreatment. The main purpose of this study is to compare the length of time that participants live without their CLL or SLL worsening between those participants who receive BGB-16673 versus the investigator's choice of treatment (idelalisib plus rituximab or bendamustine plus rituximab, or venetoclax plus rituximab).

Approximately 250 participants will be included in this study around the world. Participants will be randomly allocated to receive either BGB-16673 or the investigator's choice of treatment.

"Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website."

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CLL or SLL, requiring treatment, based on 2018 international workshop on chronic lymphocytic leukemia (iwCLL) criteria.
2. Previously received treatment for CLL/SLL with both a BTKi and a BCL2i.
3. Participants with SLL must have measurable disease by computer tomography (CT)/magnetic resonance imaging (MRI)
4. Eastern Cooperative Oncology Group (ECOG) score 0, 1, or 2
5. Adequate liver function
6. Adequate blood clotting function

Exclusion Criteria:

1. Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
2. Prior autologous stem cell transplant or chimeric antigen receptor-T cell therapy in the last 3 months
3. Known central nervous system involvement
4. Prior exposure to any BTK protein degraders
5. Active fungal, bacterial and/or viral infection requiring parenteral systemic therapy
6. Clinically significant cardiovascular disease

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-02-14 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by Independent Review Committee (IRC) | Approximately 36 Months
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by IRC using modified 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants with chronic lymphocytic leukemia (CLL) and Lugano classification for participants with small lymphocytic lymphoma (SLL).

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 36 Months
  OS is defined as time from the date of randomization to the date of death due to any cause.
Progression-Free Survival (PFS) in Participants with Prior Exposure to Noncovalent Bruton Tyrosine Kinase Inhibitor(s) (ncBTKi) by IRC | Approximately 36 Months
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by IRC using modified 2018 iwCLL for participants with prior exposure to ncBTKi.
PFS by the Investigator Assessment | Approximately 36 Months
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by the investigator using modified 2018 iwCLL criteria for participants with CLL and Lugano classification for participants with SLL
Overall Response Rate (ORR) by IRC and Investigator Assessment | Approximately 36 Months
  ORR is defined as the percentage of participants with best overall response of complete response (CR), complete response with incomplete bone marrow recovery (Cri), nodular partial remission (nPR), or partial response (PR) as assessed by the IRC or by the investigator.
Rate of Partial Response with Lymphocytosis (PR-L) or Higher Determined by IRC and by Investigator Assessment | Approximately 36 Months
  Rate of PR-L or higher is defined as the percentage of participants with a best overall response of CR, CRi, nPR, PR, or PR-L as assessed by the IRC or by the Investigator
Duration of Response (DOR) by IRC and Investigator Assessment | Approximately 36 Months
  DOR is defined as the time from initial response to disease progression or death, whichever occurs first, as assessed by the IRC or by the investigator.
Time to Next Anti-CLL/SLL Treatment (TTNT) | Approximately 36 Months
  TTNT is defined as the time from the date of randomization to the date of next anti-CLL/SLL treatment.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Approximately 36 Months
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Cancer Questionnaire -Core 30 (EORTC QLQ-C30) Global Health Status/QoL (GHS) and Physical Functioning Scales | Approximately 24 Months
  The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales(fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best). Higher scores in GHS and functional scales indicate better quality of life.
Change from baseline in EORTC Quality of Life Questionnaire - Chronic Lymphocytic Leukemia Module 17 Items (QLQ-CLL17) Symptom Burden and Physical Condition Scales | Approximately 24 Months
  The symptom burden and physical condition will be measured by QLQ-CLL17. EORTC QLQ-CLL17 comprises 17 items grouped into 3 multi-item scales: 1) symptom burden, 2) physical condition/fatigue, and 3) worries/fears about health and functioning. Each question is rated using a 4-point response scale ("not at all," "a little," "quite a bit," and "very much") and the recall period for all items is the past 7 days. The scores of each subscale are calculated based on the EORTC's protocol and then transformed to a 0 to 100 scale. Higher scores represent higher levels of symptom burden, physical condition/fatigue, or worries/fears about health and functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (94):
- United States (13):
  - St Bernards Medical Center, Jonesboro, Arkansas
  - Pih Health Whittier Hospital, Whittier, California
  - Rocky Mountain Cancer Centers (Williams) Usor, Aurora, Colorado
  - Florida Oncology and Hematology, Fort Myers, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - American Oncology Partners of Maryland Pa, Bethesda, Maryland
  - Oncology Hematology Associates, Springfield, Missouri
  - Oncology Hematology West, Pc Dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Clinical Research Alliance, Inc, Westbury, New York
  - Dayton Physician Network, Dayton, Ohio
  - Oncology Associates of Oregon Willamette Valley Cancer Center, Eugene, Oregon
  - Cancer Care Associates of York, York, Pennsylvania
  - Texas Oncology Tyler, Tyler, Texas
- Argentina (2):
  - FUNDALEU, Caba
  - Instituto Alexander Fleming (Iaf), Ciudad Autonoma Buenos Aires
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Toowoomba Hospital, Toowoomba, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Perth Blood Institute, West Perth, Western Australia
- Brazil (13):
  - CETUS, Belo Horizonte
  - Hospital Sirio Libanes Brasilia, Brasília
  - Hospital Erasto Gaertner, Curitiba
  - Centro de Ensino E Pesquisa Em Oncologia de Santa Catarina (Cepen), Florianópolis
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville
  - Complexo Hospitalar de Niteroi, Niterói
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Hospital Sao Lucas Dasa Oncologia, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro Sa, Rio de Janeiro
  - Instituto Brasileiro de Controle Do Cancer, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Germany (9):
  - Universitatsklinikum Augsburg, Augsburg
  - Praxis Am Volkspark, Berlin
  - Klinikum Chemnitz Ggmbh, Chemnitz
  - Centrum Fur Haematologie Und Onkologie Bethanien, Frankfurt am Main
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Saarland University Medical Center, Homburg
  - Invo Institut Fur Versorgungsforschung in Der Onkologie, Koblenz
  - Universitaetsklinikum Leipzig Aor, Leipzig
  - Universitatsklinikum Munster Medizinische Klinik A, Münster
- Italy (8):
  - Irccs Istituto Tumori Giovanni Paolo Ii, Bari
  - Aou Careggi, Servizio Sanitario Toscana, Florence
  - Fondazione Irccs Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Aou Maggiore Della Carita, Novara
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Ospedale Santa Maria Della Misericordia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Japan (16):
  - Nho Shikoku Cancer Center, Matsuyama, Ehime
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - Aiiku Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center, AmagasakiCity, Hyōgo
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - University Hospital, Kyoto Prefectural Univ of Medicine, KyotoShi, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Saitama Medical Center, Kawagoeshi, Saitama
  - Ntt Medical Center Tokyo, Shinagawaku, Tokyo
  - Kumamoto University Hospital, Kumamoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
- Poland (6):
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Pratia Onkologia Katowice, Katowice
  - Pratia McM Krakow, Krakow
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny Nr W Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny Im Jana Mikulicza Radeckiego We Wroclawiu, Wroclaw
- South Korea (7):
  - Dong A University Hospital, Seogu, Busan Gwang'yeogsi
  - Kyungpook National University Hospital, Junggu, Daegu Gwang'yeogsi
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, HwasunGun, Jeollanam-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Turkey (Türkiye) (5):
  - Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Gazi University, Ankara
  - Dokuz Eylul University, Balçova
  - Antalya Memorial Hospital, Dokuma
  - Sakarya Training and Research Hospital, Sakarya
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - University College Hospital, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/